CLINICAL TRIAL: NCT02701322
Title: Influence of Medical Clowning in Videofluoroscopic Examination of Pediatric Speech Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: machine malfunction and updated work rutines
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0281-15-MMC
Record Dates: First submitted 2016-02-22; First posted 2016-03-08 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Velopharyngeal Insufficiency
Keywords: Velopharyngeal Insufficiency; Fluoroscopy
MeSH Terms: conditions — Velopharyngeal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical Clown (Experimental): the study group will be accompanied by a medical clown from the arrival to the premise, through the actual examination and after exiting the exam room. The medical clown will explain about the upcoming examination and will induce a less stressed atmosphere. After the examination the clown will close the session for the patient.
  Interventions: Behavioral: Medical clown
- Control (No Intervention): The control group will do the same videofluoroscopic procedure but without a medical clown.

INTERVENTIONS:
Behavioral: Medical clown
  Arms: Medical Clown

SUMMARY:
The purpose of this study is to determine whether a participation of a medical clown in videofluoroscopic examination of pediatric speech disorder such as velopharyngeal inadequacy, improves the collaboration of the pediatric patient, the patient's and the caregivers subjective experience, and the quality of the examination (shorter exposure to radiation, shorter time at the radiology suite, more accurate parameters retrieved from the imaging results).

DETAILED DESCRIPTION:
Velopharyngeal inadequacy (VPI) results in reduced speech intelligibility and nasopharyngeal regurgitation. VPI is more common in patients who previously underwent cleft palate repair, in craniofacial syndromes such as 22q11.2 deletion syndrome, or in neuromuscular diseases. Part of the work-up sometimes includes videofluoroscopic examination of the palate's movement during speech. This procedure involves ionizing radiation and requires adequate collaboration by the examinee. The examination set-up is foreign to the child and can cause stres and anxiety which can hinder the examination's accuracy and completion. Medical clowns professionalise in stress relieve.

In this prospective controlled study, the study group will be accompanied by a medical clown from the arrival to the premise, through the actual examination and after exiting the exam room. The medical clown will explain about the upcoming examination and will induce a less stressed atmosphere. After the examination the clown will close the session for the patient.

The control group will do the same procedure but without a medical clown. Factors such as pulse, total time in the examination room, net time of exposure to radiation and quality of data will be collected for each patient. The patient (if 7 year old and up) and his caregivers will fill up after completion of the examination a short questionnaire about their experience.

The data will be collected and summarized and then a statistical analysis will be made in order to compare the study group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of velo-pharyngeal inadequacy

Exclusion Criteria:

* a patient or caregiver that did not consent to participate in the study

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
videofluoroscopy data completeness | 1 year
  The quality and completeness of radiological data that can be retrieved from the videofluoroscopy record
length of radiation exposure time | 1 year
  The length of radiation exposure time for the subject, measured in seconds

SECONDARY OUTCOMES:
Total (gross) time of examination | 1 year
  the total time the patient is in the room, measured in minutes
Subjective level of anxiety | 1 year
  the level of patient's anxiety as defined subjectively in questionnaire
Pulse | 1 year
  The difference in pulse measurement before and after the examination as an indirect assessment of level of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Yaniv Ebner, MD, Principal Investigator — Meir Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wolyniez I, Rimon A, Scolnik D, Gruber A, Tavor O, Haviv E, Glatstein M. The effect of a medical clown on pain during intravenous access in the pediatric emergency department: a randomized prospective pilot study. Clin Pediatr (Phila). 2013 Dec;52(12):1168-72. doi: 10.1177/0009922813502257. Epub 2013 Sep 11. PMID 24028842
- [Result] Goldberg A, Stauber T, Peleg O, Hanuka P, Eshayek L, Confino-Cohen R. Medical clowns ease anxiety and pain perceived by children undergoing allergy prick skin tests. Allergy. 2014 Oct;69(10):1372-9. doi: 10.1111/all.12463. Epub 2014 Aug 4. PMID 24943088